CLINICAL TRIAL: NCT07128940
Title: Biomarker pAtterns Reflecting habITual fOod iNtakE: the BARITONE Project
Acronym: BARITONE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BARITONE
Record Dates: First submitted 2025-06-26; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: food; biomarker; metabolomics; fruit and vegetables; meat; fish; plant based protein; whole grain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Meat (Experimental): All food provided for a week, including a variety of meat
  Interventions: Other: Meat vs fish; Other: Meat vs Vegetarian
- Fish (Experimental): All food provided for a week, including a variety of fish and shellfish
  Interventions: Other: Meat vs fish; Other: Fish vs Vegetarian
- Vegetarian (Experimental): All food provided for a week, diet (no fish or meat)
  Interventions: Other: Meat vs Vegetarian; Other: Fish vs Vegetarian

INTERVENTIONS:
Other: Meat vs fish — Metabolite differences: Meat vs fish
  Arms: Fish; Meat
Other: Meat vs Vegetarian — Metabolite differences: Meat vs Vegetarian
  Arms: Meat; Vegetarian
Other: Fish vs Vegetarian — Metabolite differences: Fish vs Vegetarian
  Arms: Fish; Vegetarian

SUMMARY:
The BARITONE study's overall aim is to understand how our eating habits affect our long-term health. By identifying biological traces in blood, urine and other samples - so-called biomarkers - the investigators want to be able to see what people actually eat, such as protein from different food sources as well as fruit, berries and vegetables. These biomarkers could in the future improve the possibilities to find out how dietary habits affect the risk of disease.

The investigators are targeting healthy people who are interested in participating in research on biomarkers of dietary intake. The research is divided into a cross-sectional study, where the investigators collect data on the participant's usual dietary intake, health and biological samples at the screening visit, and an cross over intervention study that involves eating three different diets (meat, fish, vegetarian) for a total of 3 weeks with one week wash-out in between.

DETAILED DESCRIPTION:
PURPOSE AND AIMS

The aims of the present project are to:

1. Identify and validate biomarker patterns of intake of the different food sources for protein, i.e., meat, fish and plant-based sources
2. Identify and validate biomarker patterns of high and low intake of the food group vegetables, fruit and berries.

Validation here includes evaluation of plausibility, robustness, and dose-response.

PROJECT DESCRIPTION Validated biomarkers are still lacking for food groups that are crucial when evaluating dietary intake, such as meat, fish and plant-based sources of protein (i.e., legumes such as lentils, peas and beans and cereal proteins such as oat- and wheat-protein); and for berries, fruits, and vegetables. For sources of protein, a well-controlled cross-over trial is needed where biomarkers of any intake of these different sources are evaluated in different biofluids. For berries, fruit and vegetables, a challenge is that no obvious control food group exists. Individuals with low consumption from this food group may instead consume any type of food. Hence, the investigators aim to evaluate biomarkers that separate consumers of low vs high intake. The investigators will follow the criteria for discovering and validating biomarkers suggested by Dragstedt et al (2018), here applied to patterns of biomarkers. The investigators will identify patterns of putative biomarkers of recent intake in biofluids in a well-controlled feeding trial (BARITONE-intervention) and develop prediction models of being a consumer/non-consumer or high/low consumer using machine learning. The robustness and dose-response of the models will be tested in data on habitual intake (BARITONE sample). Data for protein sources and berries, fruits and vegetables will be generated in the planned BARITONE-intervention trial.

Biomarker pAtterns Reflecting habITual fOod iNtakE: the BARITONE project The BARITONE project consists of two parts: 1) the BARITONE-sample (n=210) that undergoes a comprehensive baseline screening with extensive phenotyping including a 7-day weighed food diary (wk 1), and 2) the BARITONE cross-over intervention trial (n=70) where a selected group from the BARITONE-sample undergoes three dietary intervention weeks with two 7-day weighed food diaries during the two washout weeks in between.

The BARITONE-sample will be used to evaluate robustness and dose-response of putative biomarker patterns of habitual intake, because it will contain highly detailed data on habitual dietary intake and individual phenotype/metabotype. The intervention weeks of the BARITONE-trial will be used to identify putative biomarker patterns of recent intake of protein sources. Because it is a cross-over trial it allows for within-individual comparisons on metabolite reactions to dietary exposure. The wash-out periods between intervention weeks will be used to identify putative biomarker patterns of recent high or low intake of berries, fruits and vegetables, because participants will be selected based on baseline intake levels of these foods and here asked to return to their habitual diet. Hence, broad variation in intake should be represented.

The BARITONE sample for habitual diet In total, 210 healthy individuals aged 18-65 years will be invited through advertisements in media to detailed phenotyping at the laboratory of Clinical Nutrition, Gothenburg University. Procedures include a socio-demographic and lifestyle questionnaire (chronic illnesses, pharmacological treatment, physical activity, questions about menopause/timing in the menstrual cycle), a short food frequency questionnaire (FFQ), a 7-day weighed food diary and measurements of anthropometry (weight, height, body mass index, body composition by dual energy X-ray absorptiometry (DXA) or bioelectrical impedance analysis (BIA)). Biospecimens (fasting blood, spot urine; baseline stool samples) will be collected and analyzed for serum lipids, Hb, HbA1c, TSH, metabolomics including lipidomics and baseline gut microbiota.

The BARITONE cross-over intervention trial for recent intake of protein sources (Aim 1)

The BARITONE trial aims to identify metabolite patterns that can separate individuals with respect to intake of meat, fish or plant-based source of protein. From the BARITONE -sample, the investigators will select 35 participants with low intake of berries, fruit and vegetables and 35 with high intake of these same foods, to ensure a wide range of habitual intake of these foods to address Aim 2. Selection will be based on their baseline FFQ. The limit for low (<100g/day) and high intake (>400g/day) are based on the 15:th and 85:th percentile of intake data on vegetables, fruit and berries, from Riksmaten. Participants will be randomized by excel randomization function to order of trial diets by an external researcher. Blinding of participants is not possible in this diet intervention.

Intervention week diets: The diets will be identical in foods and macronutrient composition except for meat, fish or plant-based source of protein. Participants will be provided with all their food for the three trial weeks, with one week wash-out periods between the intervention periods when habitual consumption patterns should resume. Food bags will be delivered free of charge at the day before each intervention week including instructions, recipes and menus. Water will be the suggested drink. Non-sweetened drinks, coffee and tea will not be provided, but participants are allowed to consume these freely and report the intake and they should keep the consumption constant during all three intervention weeks. Alcohol will not be allowed during the intervention weeks.

The BARITONE wash-out weeks for habitual intake of berries, fruits, and vegetables (Aim 2): Detailed 7-days weighed food diaries will be collected during the two wash-out weeks among the trial participants, already selected to have low or high habitual intake of berries, fruits and vegetables. The diaries will be used to verify classification of the participants into high and low consumers. Metabolite patterns in the biofluids collected at the end of each wash-out period will be used to construct models for predicting intake of berries, fruit and vegetables, and thereafter robustness of the models will be evaluated in the BARITONE-sample.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* 18-65 years
* BMI 18.5-30 kg/m²
* Willing to consume the three diets i.e. meat, fish, and vegetarian
* Understands Swedish
* Low intake of vegetables, fruit and berries (lowest tertile of screened participants, estimated <100g day) or high intake of vegetables, fruit and berries (highest tertile of screened participants, estimated >400g day)

Exclusion Criteria:

* Pregnancy and lactation
* Diagnosis of cancer or other life threatening diseases
* Diagnosis of metabolic or food related diseases inluding diabetes, inflammatory bowel disease, hypothyroidism or celiak disease.
* Medication that influences the metabolism such as blood lipid lowering medication, insulin, etc.
* Use of drugs other than medication and alcohol
* Nicotine use (snuff, vaping and smoking)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Patterns of metabolites in plasma/serum | 1 week
  Metabolites analysed by LC-MS/GC-MS or NMR for metabolomics studies (changes in patterns of metabolites). Metabolite patterns will be compared by multivariate methods such as HDA-OPLS between the three diets. Metabolite patterns will be compared by multivariate methods such as OPLS-DA comparing high and low intake of vegetables, fruit and berries.

SECONDARY OUTCOMES:
Patterns of lipids | 1 week
  Lipids analysed by lipidomics. Changes in lipidomic patterns will be compared by multivariate methods such as HDA-OPLS between the three diets. Lipidomics patterns will be compared by multivariate methods such as OPLS-DA comparing high and low intake of vegetables, fruit and berries.
Patterns of metabolites in urine | 1 week
  Metabolites analysed by LC-MS/GC-MS or NMR for metabolomics studies (changes in patterns of metabolites). Metabolite patterns will be compared by multivariate methods such as HDA-OPLS between the three diets. Metabolite patterns will be compared by multivariate methods such as OPLS-DA comparing high and low intake of vegetables, fruit and berries.
Class disciminating metabolites in plasma/serum | 1 week
  Among the thousands of metabolites analysed by LC-MS/GC-MS or NMR for metabolomics studies a few metabolites may drive the metabolite patterns. These class discriminating metabolites (our limit is the 20 highest top-ranked variables in variable importance scores in the OPLS-HDA models) will be selected and further analysed by univariate methods.

OTHER OUTCOMES:
Fatty acid patterns in plasma | screening
  descriptive
Fatty acids in erythrocytes | screening
  descriptive
Body mass index (BMI) (kg/m2) | 1 week
  Participants should keep their weight throughout the study. BMI will be a descriptive measure or possible used for adjustment.
Fat mass (%) | baseline
  Description: Measured by dual x ray absorptiometry (DXA) or bioelectric impedance. For descriptive purposes.
Fat mass index (FMI) (kg/m2) | baseline
  Description: Measured by dual x ray absorptiometry (DXA) or bioelectric impedance. The amount of fat mass, relative to your height. For descriptive purposes.
Fat free mass index (FFMI) (kg/m2) | baseline
  Description: Measured by dual x ray absorptiometry (DXA) or bioelectric impedance. The amount of mass that is not fat, relative to your height. This includes muscle, bone, organs and connective tissue. It can be used to gauge relative muscle mass in lean individuals. For descriptive purposes.
Microbiota in feces | baseline
  Microbiota will be characterized by 16-S ribosomal gene sequencing. Descriptive for characterizing participants.
Triacylglycerides | screening
  Descriptive for characterizing participants.
Total cholesterol | screening
  Descriptive for characterizing participants.
Low density lipoprotein | screening
  Descriptive for characterizing participants.
High density lipoprotein | screening
  Descriptive for characterizing participants.
Apolipoprotein B | screening
  Descriptive for characterizing participants.
Apolipoprotein A1 | screening
  Descriptive for characterizing participants.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Not possible due to Swedish law